CLINICAL TRIAL: NCT05044741
Title: The Risk Factors for Bowel Perforation in Neonates With Hirschsprung Disease
Brief Title: Risk Factors of Perforated HSCR in Neonates
Status: Completed | Type: Observational
Sponsor: Tongji Hospital (Other)
Collaborators: Wuhan Children's Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Sponsor
Other Study IDs: Perforated HSCR
Record Dates: First submitted 2021-08-27; First posted 2021-09-16 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-08

CONDITIONS: Hirschsprung Disease; Bowel; Perforation, Fetus or Newborn
MeSH Terms: conditions — Hirschsprung Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Perforated group
  Interventions: Procedure: Emergency surgical enterostomy
- Controlled group

INTERVENTIONS:
Procedure: Emergency surgical enterostomy — Emergency surgical enterostomy
  Groups: Perforated group

SUMMARY:
Hirschsprung's disease (HSCR) is a common digestive malformation with radiographic evidence of distal bowel obstruction and clinical signs of abdominal distension, vomiting, constipation, and failure to pass meconium. Bowel perforation (perforated HSCR) is a very serious complication of HSCR, but if this occurs it is most often in the neonatal period. The current study collected information on all cases diagnosed with perforated HSCR from multi-centers in China over 10 years, the aim was to evaluate the clinical features of perforated HSCR, and investigate possible risk factors for perforated HSCR in neonates.

ELIGIBILITY:
Inclusion Criteria:

* Neonates (≤1 month age)
* Diagnosed with HSCR
* Suffered with bowel perforation

Exclusion Criteria:

* Patients complicated with suspected necrotizing enterocolitis (NEC), imperforate anus (IA), intestinal atresia, and meconium plug syndrome
* Neonates who transferred from outside participating hospitals.

Ages: 0 Days to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: -Neonates (≤1 month age) with HSCR who suffered with bowel perforation.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2006-01-01 (Actual); Primary Completion 2010-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Rate of bowel perforation in neonatal Hirschsprung disease (perforated HSCR) | 14 years
  Cases with bowel perforation in neonatal Hirschsprung disease/ total neonatal Hirschsprung disease

IPD SHARING:
Plan to Share IPD: Undecided
Until now, we do not have the plan to open individual participant data.